CLINICAL TRIAL: NCT00677924
Title: A Dose-Escalation, Randomized Phase I/II Trial of Zalutumumab - a Human Monoclonal Anti-EGF Receptor Antibody - With or Without Irinotecan Chemotherapy in Cetuximab Refractory Colorectal Cancer Patients Who Have Failed Standard Chemotherapy and Progressed During or Within 3 Months of Stopping Cetuximab-Based Therapy
Brief Title: Zalutumumab With or Without Irinotecan Chemotherapy in Cetuximab-Refractory Colorectal Cancer
Acronym: GEN206
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to changes in portfolio review
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEN206
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Neoplasms; Colorectal Tumors; Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zalutumumab 8 mg/kg (Experimental): Zalutumumab in combination with Irinotecan
  Interventions: Drug: Zalutumumab
- Zalutumumab 16 mg/kg (Experimental): Zalutumumab in combination with Irinotecan
  Interventions: Drug: Zalutumumab

INTERVENTIONS:
Drug: Zalutumumab — Solution for infusion
  Other Names: HuMax-EGFr

SUMMARY:
The purpose of this trial is to determine the safety and efficacy of Zalutumumab alone or in combination with Irinotecan for the treatment of patients with Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females age ≥ 18 years
2. Confirmed diagnosis of CRC
3. Documented disease progression
4. Failure and/or intolerance to standard chemotherapy

Exclusion Criteria:

1. Prior treatment with anti-EGFR antibodies other than cetuximab
2. Expected survival < 3 months
3. Clinical significant cardiac disease and/or uncontrolled medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Aladdin, ICTM, Study Director — Genmab
Locations (3):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Hospital Erasme, Brussels
  - St-Luc University Hospital, Brussels

REFERENCES:
- [Result] Mano M, Hendlisz A, Machiels JP, Ehrnrooth E, Aladdin H, Van Laethem JL. Phase I trial of zalutumumab and irinotecan in metastatic colorectal cancer patients who have failed irinotecan and cetuximab based therapy. J Clin Oncol 27 2009 (suppl;abstr e15028)

RESULTS

PARTICIPANT FLOW:
Groups:
- Zalatumumab 8 mg/kg: Participants received zalutumumab 8 milligrams per kilogram (mg/kg) intravenously once weekly in combination with irinotecan 180 milligrams per meter square (mg/m^2) every 2 weeks up to 10 months.
- Zalutumumab 16 mg/kg: Participants received zalutumumab 16 mg/kg intravenously once weekly in combination with irinotecan 180 mg/m^2 every 2 weeks up to 10 months.
Period: Overall Study
Arm/Group | Zalatumumab 8 mg/kg | Zalutumumab 16 mg/kg
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zalatumumab 8 mg/kg: Participants received zalutumumab 8 mg/kg intravenously once weekly in combination with irinotecan 180 mg/m^2 every 2 weeks up to 10 months.
- Total: Total of all reporting groups
Arm/Group | Zalatumumab 8 mg/kg | Zalutumumab 16 mg/kg | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 1 | 1 | 2
Age, Continuous [Median (Full Range); unit: years] | 61 [57 to 66] | 61 [33 to 76] | 61 [33 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Belgium | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From first dose up to follow-up (up to approximately 1 year)
Population: All participants who had been exposed to zalutumumab or irinotecan, irrespective of their compliance to the planned course of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Zalatumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 3 | 6
Participants | 3 | 5

2. Secondary Outcome: Number of Participants With Best Overall Tumour Response (BOR)
Description: The BOR defined as the best response recorded from the start of treatment until disease progression or recurrence per RECIST criteria. Complete response (CR) defined as the disappearance of all target lesions. Partial response (PR) defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Progressive disease (PD) defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, or the appearance of one or more new lesions since the prior scan. Stable disease (SD) defined as responses not fulfilling CR, PR or PD.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Zalatumumab 8 mg/kg | Zalutumumab 16 mg/kg
Number analyzed (Participants) | 3 | 6
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 3 | 4
  Progressive Disease | 0 | 2

ADVERSE EVENTS:
Time Frame: From first dose up to follow-up (up to approximately 1 year)
Arm/Group | Zalatumumab 8 mg/kg | Zalutumumab 16 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalatumumab 8 mg/kg (N=3) | Zalutumumab 16 mg/kg (N=6)
Disease progression (General disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalatumumab 8 mg/kg (N=3) | Zalutumumab 16 mg/kg (N=6)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Fatigue (General disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Disease progression (General disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1)
Myalgia (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The trial was prematurely closed when 9 out of 97 patients were enrolled. The trial design was originally divided in two parts. Patient allocation was terminated before Part 2 was started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The site and the PI may be required to withhold the publication for up to 90 days. Subject to a reasoned request from the sponsor, the publication may be further delayed for a period up to 6 months from the date of first submission to the sponsor.

The sponsor has the right to require deletion of any trade secret, proprietary, or confidential information supplied by the sponsor to the site or the PI. The sponsor shall not otherwise have the right to censor publications.